CLINICAL TRIAL: NCT00238953
Title: A Prospective, Open Label Protocol to Assess the Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in de Novo Kidney Transplant Recipients
Brief Title: Efficacy and Safety of Enteric-coated Mycophenolate Sodium (EC-MPS) in de Novo Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080APL01
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Renal Transplantation
Keywords: Kidney transplantation; enteric-coated mycophenolate sodium

ARMS (1):
- EC MPS (Experimental)
  Interventions: Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
Clinical trial for the novo transplant recipients, which aims to assess tolerability and safety and clinical outcomes of EC-MPS in combination with cyclosporine microemulsion (CsA-ME) with or without steroids in a population of kidney transplant recipients.

ELIGIBILITY:
Inclusion criteria:

* Male and females aged 18 to 75
* Recipients of cadaveric, living unrelated or living related kidney transplant, treated with CsA-ME, with or without corticosteroids, as primary immunosuppression

Exclusion criteria:

* Multi-organ recipients (e.g. kidney and pancreas) or previous transplant with any organ, other than kidney.
* Patients with any known hypersensitivity to MPA, EC-MPS or other components of the formulation (e.g. lactose).
* Patients with thrombocytopenia (< 75,000/mm3), with an absolute neutrophil count of < 1,500/mm3, and/or leukocytopenia (< 2,500/mm3), and/or hemoglobin < 6 g/dL at Screening or Baseline.

Other inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
6 Month evaluation
patient and graft survival
acute rejection (suspected or biopsy confirmed)
graft function (serum creatinine, calculated creatinine clearance and glomerular filtration rate),
infections, adverse events, serious adverse events.

SECONDARY OUTCOMES:
Influence of parameters: demography, medical conditions, complications post transplantation on main clinical outcomes. 6 month evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Wyzgal J, Niemczyk M, Ziolkowski J, Durlik M, Wiecek A. Results of a 6-month, multicenter, open-label, prospective study concerning efficacy and safety of mycophenolate sodium in de novo kidney transplant recipients. Transplant Proc. 2007 Nov;39(9):2730-2. doi: 10.1016/j.transproceed.2007.08.071. PMID 18021971